CLINICAL TRIAL: NCT03209934
Title: Daptomycin > 6 mg/kg/Day as Salvage Therapy in Patients With Complex Bone and Joint Infection: Cohort Study in a Regionalreference Center
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0465
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Bone and Joint Infection; Treated by Daptomycin
Keywords: Bone and Joint Infection; Daptomycin; Eosinophilic pneumonia
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The choice of antimicrobial therapy to treat complex bone and joint infections (BJI) is challenging, requiring consideration of: (i) the problem of bone diffusion; (ii) the necessity of using antimicrobials active against bacterial biofilms; (iii) the growing incidence of antibiotic resistance; and (iv) the high risk of severe adverse events (SAE) in response to first-line antimicrobials in these patients.

Consequently, off-label use of recently developed antimicrobials, such as daptomycin, is frequently required as salvage therapy in complex BJI. Even if daptomycin does not have approval for the treatment of BJI, the Infectious Diseases Society of America guidelines propose this antibiotic as alternative therapy for prosthetic joint infection. The recommended dose is 6 mg/kg/d, whereas recent data support the use of higher doses in these patients as bone penetration of daptomycin is limited.

The present cohort study aimed to assess the safety and efficacy of prolonged high-dose (>6 mg/kg/d) daptomycin salvage therapy in patients with complex BJI.

ELIGIBILITY:
Inclusion Criteria:

* patients having BJI treated by daptomycin at >6 mg/kg/d

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who received daptomycin >6 mg/kg/d as an alternative therapy for complex BJI from January 2011 to July 2013 in a French regional reference center.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Measure of daptomycin through plasma concentration (Cmin) | 300 days
  The approximal maximal treatment duration is 300 days. Daptomycin trough plasma concentration (Cmin) is determined monthly to detect any patients with daptomycin trough levels (Cmin) over 24 mg/L. Cmin is determined 24 h after daptomycin injection (just before reinjection, if performed) using a validated HPLC process developed in the laboratory and a diode array UV detector.
  Cmin > 24 mg/L was considered an overdose, as the risk of high CPK levels (with or without symptoms of myopathy) is greater above this threshold